CLINICAL TRIAL: NCT01124864
Title: A Phase II, Multi-center, Open-label Study of AUY922 Administered IV on a Once-weekly Schedule in Patients With Advanced Non-small-cell Lung Cancer Who Have Received at Least Two Lines of Prior Chemotherapy
Brief Title: A Study of AUY922 in Non-small-cell Lung Cancer Patients Who Have Received Previous Two Lines of Chemotherapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAUY922A2206; 2010-020116-11 (EudraCT Number)
Record Dates: First submitted 2010-05-14; First posted 2010-05-17 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Non-small-cell lung cancer; HSP90; 2nd to 3rd line treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- EGFR mutant patients (Experimental): Patients with EGFR activating mutation tumors (Note: These patients must have progressed on one prior EGFR TKI containing regimen unless they have documented T790M activating mutation). Patients received AUY922 at 70 mg/m^2 weekly infusions.
  Interventions: Drug: AUY922
- Kras mutant patients (Experimental): Patients with KRAS mutant tumors. Patients received AUY922 at 70 mg/m^2 weekly infusions.
  Interventions: Drug: AUY922
- EGFR and Kras wild type patients (Experimental): Patients exhibiting both mutations were stratified to the KRAS mutation stratum. Patients received AUY922 at 70 mg/m^2 weekly infusions.
  Interventions: Drug: AUY922
- Patients with EML4-ALK translocation (Experimental): Patients with NSCLC who have tumors with an inversion in the short arm of chromosome 2 that results in the fusion of the echinoderm microtubule-associated protein-like 4 (EML4) gene with the ALK gene leading to the production of an EML4-ALK fusion tyrosine kinase. ALK is a transmembrane protein, which has a kinase domain and is not usually expressed in the lung. EML4 mediate ligand-independent dimerization, and therefore constitutive activity of the ALK tyrosine kinase domain. Patients received AUY922 at 70 mg/m^2 weekly infusions.
  Interventions: Drug: AUY922
- Modified EGFR mutant patients (Experimental): The modified EGFR stratum was defined as patients less heavily pretreated who had received one or two lines of prior therapy, with a documented response to a EGFR tyrosine kinase inhibitor (TKI) (complete response (CR), partial response (PR) or stable disease (SD) for ≥ 6 months), unless the patient had de novo resistance to EGFR TKI. Patients received AUY922 at 70 mg/m^2 weekly infusions.
  Interventions: Drug: AUY922

INTERVENTIONS:
Drug: AUY922 — AUY922 was supplied in individual 10 mL amber colored glass ampoules containing 10 mL of a 5 mg/mL active drug substance in 5% aqueous glucose solution. AUY922 was administered intravenously (i.v.) weekly at 70 mg/m2.

SUMMARY:
This study will assess the efficacy of AUY922, when administered weekly at 70 mg/m2, in adult patients with advanced Non-small-cell Lung Cancer (NSCLC), who have received at least two prior lines of chemotherapy. Patients will be retrospectively, and prospectively, stratified based on their molecular tumor etiology. The following strata was assigned: Patients with Epidermal growth factor receptor (EGFR) activating mutations, Patients with Kirstin Raus sarcoma virus (KRAS) activating mutations, Patients with EML4-ALK (anaplastic lymphoma kinase) translocations and patients that were both EGFR and Kras wild type.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced (stage IIIB or stage IV) NSCLC who have received at least two prior lines of treatment. Patients who, in the investigators opinion, are deemed unsuitable for the standard 2nd line chemotherapy will be eligible for protocol participation. One of the prior lines must have included a platinum agent. Prior treatment with a platinum agent is not a requirement for EGFR mutant patients and patients with EML4-ALK translocations
* Patients enrolled to the fifth stratum, modified EGFR mutant, must have documented prior response to EGFR TKI as defined by CR, PR or SD for 6 months or greater unless patient has de novo resistance to EGFR TKI (e.g. exon 20 insertions.)
* All patients must have at least one measurable lesion as defined by RECIST criteria. Previously irradiated lesions are not measurable unless the lesion is new or has demonstrated clear progression after radiation
* World Health Organization (WHO) performance status ≤ 2. For patients enrolled to the fifth stratum, modified EGFR mutant, World Health Organization (WHO) performance status ≤ 1
* Patients enrolled to the fifth stratum, modified EGFR mutant, must be willing and suitable to undergo fresh baseline biopsy prior to study treatment (unless patient had recent biopsy after EGFR TKI progression that concluded resistance to EGFR TKI.)
* Hematologic:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L.
  * Hemoglobin (Hgb) ≥ 9 g/dl.
  * Platelets (plt) ≥ 100 x 109/L.

Biochemistry:

* Total calcium (corrected for serum albumin) within normal limits or correctable with supplements.
* Magnesium within lower normal limits or correctable with supplements.

Adequate liver function defined as:

* AST/SGOT and ALT/SGPT ≤ 3.0 x Upper limit of Normal (ULN) or ≤ 5.0 x ULN if liver metastasis are present.
* Serum bilirubin ≤ 1.5 x ULN.
* Serum albumin > 2.5 g/dL.
* Serum creatinine ≤ 1.5 x ULN or 24 hour clearance ≥ 50 mL/min.

Exclusion Criteria:

* Patients who have received more than four lines of prior treatment. Exception: Patients enrolled to the fifth stratum, modified EGFR mutant, must not have received more than two prior lines of therapy. Chemotherapy administered as adjuvant treatment more than six months prior to study enrollment is not considered a prior line of therapy for purposes of this study.
* Patients with a history of CNS metastasis. Note: Patients without clinical signs and symptoms of CNS involvement are not required to have MRI of the brain. Exception: Patients with treated brain metastases who are asymptomatic, who has discontinued corticosteroids, and who have been clinically stable for one month will be eligible for protocol participation. This exception is not valid for patients enrolled to the fifth stratum, modified EGFR mutant. These patients must not have CNS involvement.
* Prior anti-neoplastic treatment with any HSP90 or HDAC inhibitor compound.
* Patients must not have received:

  * any systemic anti-cancer treatment or radiotherapy within 4 weeks prior to first dose of study treatment and should have recovered to baseline or less than Grade 1 from toxicities of such therapy prior to the first dose of study treatment
  * 2 weeks for palliative radiotherapy to bones, 6 weeks for nitrosoureas and mitomycin
  * 4 weeks for monoclonal antibodies
  * and ≤5 half-life of the agent or active metabolites [if any] for continuous systemic anti-cancer treatment or investigational
* Patients who do not have either an archival tumor sample available or are unwilling to have a fresh tumor sample collected at baseline.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2010-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (4):
  - University of California at Los Angeles UCLA - Santa Monica, Los Angeles, California
  - Maryland Oncology Hematology, P.A. Dept. of Assoc. Onc/Hem, Rockville, Maryland
  - Dana Farber Cancer Institute DFCI, Boston, Massachusetts
  - St. Luke's Hospital and Health Network St Luke's, Bethlehem, Pennsylvania
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Montreal, Quebec
- France (3):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Villejuif
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Oldenburg
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (2):
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
- Novartis Investigative Site, Izmir, Turkey, Turkey (Türkiye)

REFERENCES:
- [Derived] Felip E, Barlesi F, Besse B, Chu Q, Gandhi L, Kim SW, Carcereny E, Sequist LV, Brunsvig P, Chouaid C, Smit EF, Groen HJM, Kim DW, Park K, Avsar E, Szpakowski S, Akimov M, Garon EB. Phase 2 Study of the HSP-90 Inhibitor AUY922 in Previously Treated and Molecularly Defined Patients with Advanced Non-Small Cell Lung Cancer. J Thorac Oncol. 2018 Apr;13(4):576-584. doi: 10.1016/j.jtho.2017.11.131. Epub 2017 Dec 13. PMID 29247830

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two patients who were ongoing at the data cut-off of 30-Jul-2013 are considered as 'completed' in this study.
Groups:
- FG005: For some patients, it was not possible to determine their genotype, and hence their stratum membership could not be determined. Patients received AUY922 at 70 mg/m^2 weekly infusions.
Period: Overall Study
Arm/Group | Kras Mutant Patients | EGFR Mutant Patients | EGFR and Kras Wild Type Patients | Patients With EML4-ALK Translocation | Modified EGFR Mutant Patients | FG005
Started | 28 | 35 | 34 | 22 | 31 | 3
Completed | 0 | 0 | 0 | 1 (1 patient ongoing at time of data cut-off 30-Jul-2013) | 1 (1 patient ongoing at time of data cut-off 30-Jul-2013) | 0
Not Completed | 28 | 35 | 34 | 21 | 30 | 3
Not completed — Follow up phase competed as per protocol | 18 | 22 | 24 | 18 | 26 | 2
Not completed — Death | 6 | 9 | 6 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 4 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all patients who received at least one dose of AUY922.
Groups:
- Unknown: For some patients, it was not possible to determine their genotype, and hence their stratum membership could not be determined. Patients received AUY922 at 70 mg/m^2 weekly infusions.
- Total: Total of all reporting groups
Arm/Group | Kras Mutant Patients | EGFR Mutant Patients | EGFR and Kras Wild Type Patients | Patients With EML4-ALK Translocation | Modified EGFR Mutant Patients | Unknown | Total
Number analyzed (Participants) | 28 | 35 | 34 | 22 | 31 | 3 | 153
Age, Customized [Number; unit: Participants]
  < 65 years | 20 | 21 | 23 | 18 | 25 | 1 | 108
  >= 65 years | 8 | 14 | 11 | 4 | 6 | 2 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 25 | 18 | 15 | 19 | 0 | 88
  Male | 17 | 10 | 16 | 7 | 12 | 3 | 65
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 25 | 25 | 23 | 16 | 16 | 2 | 107
  Black | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 10 | 9 | 6 | 13 | 1 | 41
  Other | 1 | 0 | 1 | 0 | 2 | 0 | 4
Height [Mean (Standard Deviation); unit: cm] | 170.5 (9.94) | 163.0 (6.63) | 165.8 (10.32) | 164.9 (9.80) | 163.9 (8.93) | 173.0 (14.73) | 165.7 (9.49)
Weight [Mean (Standard Deviation); unit: kg] | 74.5 (16.22) | 64.0 (12.05) | 68.4 (13.49) | 60.5 (12.30) | 67.1 (11.02) | 76.6 (15.75) | 67.3 (13.70)
Weight category [Number; unit: Participants]
  < 55 kg | 4 | 10 | 4 | 10 | 4 | 0 | 32
  55 - <75 kg | 13 | 19 | 21 | 9 | 20 | 2 | 84
  >= 75 kg | 11 | 6 | 9 | 3 | 7 | 1 | 37
Body surface area [Mean (Standard Deviation); unit: m^2] | 1.9 (0.23) | 1.7 (0.18) | 1.8 (0.21) | 1.7 (0.20) | 1.8 (0.18) | 1.9 (0.27) | 1.8 (0.21)
Percentage of LVEF (left ventricular ejection fraction) [Mean (Standard Deviation); unit: Percentage of LVEF] | 63.2 (8.92) | 66.9 (7.63) | 66.2 (9.27) | 69.5 (8.68) | 65.4 (7.64) | 69.0 (10.54) | 66.2 (8.51)
WHO Performance status [Number; unit: Participants] — Who Performance status:
  0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work
  2. Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours
  Participants
    Who Performance status: 0 | 10 | 13 | 10 | 9 | 11 | 1 | 54
    Who Performance status: 1 | 18 | 19 | 21 | 11 | 20 | 2 | 91
    Who Performance status: 2 | 0 | 3 | 3 | 2 | 0 | 0 | 8
Smoking status [Number; unit: Participants]
  Current smoker | 3 | 1 | 2 | 2 | 1 | 1 | 10
  Ex-smoker | 21 | 12 | 18 | 5 | 16 | 0 | 72
  Never smoked | 4 | 22 | 14 | 15 | 14 | 2 | 71
Time since smoking cessation [Mean (Standard Deviation); unit: months] | 59.0 (80.65) | 176.6 (15.04) | 180.3 (120.88) | NA (NA) — No patients were analyzed in this group. | 340.4 (179.18) | NA (NA) — No patients were analyzed in this group. | 152.4 (142.22)

OUTCOME MEASURES:

1. Primary Outcome: Response Assessment by Study Stratum - Per Investigator Assessment
Description: The primary endpoint of the study was the investigator assessment of efficacy at 18 weeks in terms of response complete response (CR)/partial response (PR), stable disease (SD), or non clinical benefit (NCB) as assessed by response evaluation criteriain solid tumors (RECIST) version 1.0. ORR = patients with confirmed complete or partial response. Stable disease at 18 weeks = patients without response and with no assessment of progressive disease up to 18 weeks, but with an assessment of stable disease or better either within 2 weeks prior to the 18 week time point, or at the next non-missing assessment after the 18 week time point. No clinical benefit = all other patients.
Time Frame: 18 weeks
Population: The Full Analysis Set (FAS) consisted of all patients who received at least one dose of AUY922.
Measure: Number; unit: Participants
Arm/Group | Kras Mutant Patients | EGFR Mutant Patients | EGFR and Kras Wild Type Patients | Patients With EML4-ALK Translocation | Modified EGFR Mutant Patients | Unknown
Number analyzed (Participants) | 28 | 35 | 34 | 22 | 31 | 3
Participants
  Overall respose rate (ORR) | 0 | 6 | 3 | 7 | 3 | 1
  Stable disease for ≥18 weeks | 2 | 3 | 3 | 2 | 7 | 0
  No clinical benefit | 26 | 26 | 28 | 13 | 21 | 2

2. Secondary Outcome: Overall Survival Rate Using Kaplan Meier Estimates - Per Investigator Radiological Review
Description: Overall survival (OS) is defined as the time from date of randomization/start of treatment to date of death due to any cause. If a patient is not known to have died, survival was censored at the date of last contact.
Time Frame: Week 12, Week 18
Population: The Full Analysis Set (FAS) consisted of all patients who received at least one dose of AUY922.
Measure: Number; unit: Percentage of participants
Arm/Group | Kras Mutant Patients | EGFR Mutant Patients | EGFR and Kras Wild Type Patients | Patients With EML4-ALK Translocation | Modified EGFR Mutant Patients | Unknown
Number analyzed (Participants) | 28 | 35 | 34 | 22 | 31 | 3
Percentage of participants
  12 weeks | 68.7 [47.0 to 83.0] | 77.0 [59.3 to 8708] | 78.6 [60.2 to 89.2] | 90.7 [67.6 to 97.6] | 96.7 [78.6 to 99.5] | 66.7 [5.4 to 94.5]
  18 weeks | 55.9 [34.4 to 72.8] | 74.1 [56.1 to 85.6] | 72.3 [53.5 to 84.5] | 71.6 [47.4 to 86.1] | 93.3 [75.9 to 98.3] | 33.3 [0.9 to 77.4]

3. Secondary Outcome: Progression Free Survival (PFS) Rate as Per Investigator Using Kaplan Meier Estimates - Per Investigator Radiological Review
Description: Progression-free survival (PFS) is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient did not have an event, progression-free survival was censored at the date of last adequate tumor assessment. A Novartis modified response evaluation criteria in solid tumors RECIST 1.1 criteria was applied to CT/MRI imaging data when assessing any responses to AUY922 treatment. All images were evaluated locally by the investigator. All complete or partial responses were confirmed by a second assessment at least 4 weeks later.
Time Frame: Week 12, Week 18
Population: The Full Analysis Set (FAS) consisted of all patients who received at least one dose of AUY922.
Measure: Number; unit: Percentage of participants
Arm/Group | Kras Mutant Patients | EGFR Mutant Patients | EGFR and Kras Wild Type Patients | Patients With EML4-ALK Translocation | Modified EGFR Mutant Patients | Unknown
Number analyzed (Participants) | 28 | 35 | 34 | 22 | 31 | 3
Percentage of participants
  12 weeks | 31.5 [14.9 to 49.6] | 44.4 [27.0 to 60.5] | 31.5 [16.3 to 47.9] | 45.5 [24.4 to 64.3] | 56.4 [36.9 to 72.0] | 33.3 [0.9 to 77.4]
  18 weeks | 9.0 [1.6 to 24.6] | 27.7 [13.5 to 43.9] | 24.0 [10.6 to 40.3] | 36.4 [17.4 to 55.7] | 37.8 [20.4 to 55.1] | 33.3 [0.9 to 77.4]

4. Secondary Outcome: Pharmacokinetics (PK) of Plasma Concentration of AUY922 and Its Metabolite BJP762: AUCinf
Description: Summary of PK parameters for all patients one hour post 70 mg/m2 AUY922 infusion for area under the curve infinity. There are discrepancies between sample numbers and study population because PK samples were not collected from all study subjects and thus were not analyzed.
Time Frame: 1 hour after infusion
Population: PK analysis subset - All patients who received at least one dose of AUY922 in Cycle 1 and had at least one measurable post-dose AUY922 concentration.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- AUY922: AUY922 Plasma Concentration
- BJP762: AUY Metabolite
Arm/Group | AUY922 | BJP762
Number analyzed (Participants) | 119 | 117
h*ng/mL | 2101.27 (990.320) | 13963.07 (13006.537)

5. Secondary Outcome: Pharmacokinetics (PK) of Plasma Concentration of AUY922 and Its Metabolite BJP762: AUClast
Description: Summary of PK parameters for all patients one hour post 70 mg/m2 AUY922 infusion for area under the curve last. There are discrepancies between sample numbers and study population because PK samples were not collected from all study subjects and thus were not analyzed.
Time Frame: 1 hour after infusion
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | AUY922 | BJP762
Number analyzed (Participants) | 139 | 142
h*ng/mL | 1997.04 (894.903) | 12496.75 (12035.525)

6. Secondary Outcome: Pharmacokinetics (PK) of Plasma Concentration of AUY922 and Its Metabolite BJP762: Cmax
Description: Summary of PK parameters for all patients one hour post 70 mg/m2 AUY922 infusion for concentration max. There are discrepancies between sample numbers and study population because PK samples were not collected from all study subjects and thus were not analyzed.
Time Frame: 1 hour after infusion
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AUY922 | BJP762
Number analyzed (Participants) | 144 | 144
ng/mL | 1130.59 (705.177) | 2332.86 (1377.350)

ADVERSE EVENTS:
Groups:
- KRAS Mutant: Patients with KRAS mutant tumors. Patients received AUY922 at 70 mg/m^2 weekly infusions.
- EGFR Mutant: Patients with EGFR activating mutation tumors (Note: These patients must have progressed on one prior EGFR TKI containing regimen unless they have documented T790M activating mutation). Patients received AUY922 at 70 mg/m^2 weekly infusions.
- KRAS and EGFR Wild Type: Patients exhibiting both mutations were stratified to the KRAS mutation stratum. Patients received AUY922 at 70 mg/m^2 weekly infusions.
- EML4-ALK Translocation: Patients with NSCLC who have tumors with an inversion in the short arm of chromosome 2 that results in the fusion of the echinoderm microtubule-associated protein-like 4 (EML4) gene with the ALK gene leading to the production of an EML4-ALK fusion tyrosine kinase. ALK is a transmembrane protein, which has a kinase domain and is not usually expressed in the lung. EML4 mediate ligand-independent dimerization, and therefore constitutive activity of the ALK tyrosine kinase domain. Patients received AUY922 at 70 mg/m^2 weekly infusions.
- Modified EGFR Mutant: The modified EGFR stratum was defined as patients less heavily pretreated who had received one or two lines of prior therapy, with a documented response to a EGFR tyrosine kinase inhibitor (TKI) (complete response (CR), partial response (PR) or stable disease (SD) for ≥ 6 months), unless the patient had de novo resistance to EGFR TKI.Patients received AUY922 at 70 mg/m^2 weekly infusions.
- EG005: For some patients, it was not possible to determine their genotype, and hence their stratum membership could not be determined. Patients received AUY922 at 70 mg/m^2 weekly infusions.
Arm/Group | KRAS Mutant | EGFR Mutant | KRAS and EGFR Wild Type | EML4-ALK Translocation | Modified EGFR Mutant | EG005
Serious Adverse Events (participants affected / at risk) | 17/28 | 18/35 | 22/34 | 6/22 | 11/31 | 2/3
Other Adverse Events (participants affected / at risk) | 28/28 | 35/35 | 33/34 | 22/22 | 31/31 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KRAS Mutant (N=28) | EGFR Mutant (N=35) | KRAS and EGFR Wild Type (N=34) | EML4-ALK Translocation (N=22) | Modified EGFR Mutant (N=31) | EG005 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 2 | 0 | 0 | 0
Bundle Branch Block Right (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Night Blindness (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal Fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 1 | 0
General Physical Health Deterioration (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 2 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Klebsiella Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Perirectal Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 1 | 1 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0
Failure To Thrive (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Fluid Intake Reduced (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Balance Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Brain Compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nervous System Disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vocal Cord Paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 3 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KRAS Mutant (N=28) | EGFR Mutant (N=35) | KRAS and EGFR Wild Type (N=34) | EML4-ALK Translocation (N=22) | Modified EGFR Mutant (N=31) | EG005 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 5 | 3 | 4 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 1 | 1 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 2 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 2 | 2 | 1 | 0
Accommodation Disorder (Eye disorders) | 1 | 2 | 2 | 2 | 5 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 0
Cataract Subcapsular (Eye disorders) | 1 | 0 | 2 | 0 | 0 | 0
Colour Blindness Acquired (Eye disorders) | 0 | 3 | 2 | 5 | 4 | 1
Dry Eye (Eye disorders) | 2 | 0 | 1 | 2 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 1 | 0 | 2 | 0
Lacrimation Increased (Eye disorders) | 0 | 2 | 0 | 0 | 1 | 0
Loss Of Visual Contrast Sensitivity (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0
Night Blindness (Eye disorders) | 3 | 10 | 6 | 5 | 10 | 1
Ocular Toxicity (Eye disorders) | 4 | 4 | 1 | 3 | 3 | 1
Photophobia (Eye disorders) | 3 | 2 | 5 | 0 | 2 | 0
Photopsia (Eye disorders) | 3 | 5 | 10 | 10 | 6 | 0
Retinal Disorder (Eye disorders) | 1 | 3 | 1 | 5 | 7 | 0
Vision Blurred (Eye disorders) | 5 | 6 | 7 | 6 | 6 | 0
Visual Acuity Reduced (Eye disorders) | 1 | 6 | 7 | 7 | 5 | 0
Visual Impairment (Eye disorders) | 6 | 8 | 3 | 6 | 7 | 0
Vitreous Floaters (Eye disorders) | 1 | 3 | 1 | 1 | 2 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 5 | 5 | 4 | 6 | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 3 | 2 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 6 | 6 | 5 | 5 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 25 | 23 | 25 | 17 | 24 | 3
Dry Mouth (Gastrointestinal disorders) | 5 | 4 | 6 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 4 | 3 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 16 | 19 | 13 | 11 | 12 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 13 | 13 | 4 | 9 | 4 | 2
Asthenia (General disorders) | 13 | 14 | 10 | 10 | 5 | 1
Catheter Site Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Chest Pain (General disorders) | 1 | 2 | 0 | 4 | 0 | 1
Fatigue (General disorders) | 7 | 9 | 13 | 3 | 15 | 0
Gait Disturbance (General disorders) | 0 | 2 | 2 | 2 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 2 | 2 | 1 | 0
Oedema Peripheral (General disorders) | 2 | 2 | 1 | 3 | 3 | 0
Pain (General disorders) | 1 | 2 | 6 | 0 | 1 | 1
Pyrexia (General disorders) | 5 | 3 | 4 | 6 | 4 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 4 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 1 | 2 | 4 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 2 | 1 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 1 | 2 | 2 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 4 | 1 | 1 | 3 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1
C-Reactive Protein Increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 2 | 1 | 0 | 3 | 0
Heart Rate Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hypophonesis (Investigations) | 0 | 0 | 1 | 2 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Weight Decreased (Investigations) | 4 | 1 | 3 | 1 | 4 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 17 | 15 | 12 | 8 | 10 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 3 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 2 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 5 | 8 | 3 | 7 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 3 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 3 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 1 | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5 | 1 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 5 | 6 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 1 | 2 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 4 | 1 | 1 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Balance Disorder (Nervous system disorders) | 1 | 0 | 0 | 1 | 3 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 1 | 3 | 1
Dysgeusia (Nervous system disorders) | 2 | 1 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 8 | 8 | 8 | 14 | 13 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 2 | 2 | 0
Memory Impairment (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 3 | 1 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 3 | 3 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 2 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 2 | 3 | 2 | 2 | 0
Depressed Mood (Psychiatric disorders) | 0 | 1 | 2 | 2 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 6 | 5 | 4 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 2 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 9 | 7 | 8 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 9 | 2 | 2 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 3 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 2 | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 7 | 2 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 4 | 0
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 1 | 0 | 1 | 2 | 1 | 0
Hypertension (Vascular disorders) | 0 | 4 | 3 | 3 | 5 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.